CLINICAL TRIAL: NCT01216709
Title: Iron Absorption From Iron-fortified Infant Formula and Iron Drops in Infants (MJAU-studien)
Brief Title: Iron Absorption From Infant Formula and Iron Drops in Infants (MJAU-studien)
Acronym: MJAU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Umeå University (Other)
Collaborators: Swiss Federal Institute of Technology (Other); University of California, Davis (Other)
Responsible Party: Principal Investigator, Magnus Domellöf, MD, PhD, Umeå University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: Iron absorption in infants
Record Dates: First submitted 2010-10-06; First posted 2010-10-07 (Estimated); Last update posted 2020-03-26 (Actual); Status verified 2020-03

CONDITIONS: Infant; Dietary Supplements; Food, Fortified
Keywords: Infant; Dietary Supplements; Food, Fortified; Iron Absorption
MeSH Terms: interventions — ferrous sulfate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- iron drops (Experimental)
  Interventions: Dietary Supplement: ferrous sulfate
- iron-fortified formula (2.3 mg iron/L) (Experimental)
  Interventions: Other: iron-fortified infant formula (2.3 mg iron/L)
- iron-fortified formula (12.4 mg iron /L) (Experimental)
  Interventions: Other: iron-fortified infant formula (12.4 mg iron/L)

INTERVENTIONS:
Dietary Supplement: ferrous sulfate — 6.3 mg iron from iron drops and 0.3 mg iron from infant formula with no added iron (0.5 mg iron/L) for 45 days
  Arms: iron drops
Other: iron-fortified infant formula (12.4 mg iron/L) — 6.6 mg iron from iron-fortified infant formula (12.4 mg iron/L) for 45 days
  Arms: iron-fortified formula (12.4 mg iron /L)
Other: iron-fortified infant formula (2.3 mg iron/L) — 1.2 mg iron from iron-fortified infant formula (2.3 mg iron/L) for 45 days
  Arms: iron-fortified formula (2.3 mg iron/L)

SUMMARY:
Iron deficiency (ID) affects up to 25% of Swedish infants and severe ID is associated with cognitive and behavioral problems. To avoid this, iron supplements or iron-fortified infant foods are recommended for infants. However, the optimal iron dose and mode of delivery have not yet been established. This is a concern as excessive iron intake may impair growth and increase morbidity in iron-sufficient infants. Previous studies have suggested that iron-fortified foods may have different effects than iron supplements. In this study, the investigators will investigate whether the mode of iron administration (supplementation vs. fortification) and the amount consumed (high intakes vs. low intakes) affect iron absorption, iron utilization, and zinc absorption in healthy term non-iron-deficient 6-month-old infants.

ELIGIBILITY:
Inclusion Criteria:

* 6-7 months of age at the start of intervention
* healthy at enrollment
* full-term (>37 gestational weeks at birth)
* birth weight >2500 g
* predominantly bottle-fed at recruitment

Exclusion Criteria:

* iron deficiency at enrollment
* previous or current use of iron supplements

Ages: 6 Months to 7 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 72 (Actual)
Dates: Start 2010-10 (Actual); Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
iron absorption | 1 month after enrollment

SECONDARY OUTCOMES:
indicators of iron metabolism, growth, and oxidative stress | 1 month and 1.5 months after enrollment
zinc absorption | 1 month after enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Magnus Domellöf, MD, PhD, Principal Investigator — Umeå University
Locations (1):
- Department of Clinical Sciences, Pediatrics, Umeå University Hospital, Umeå, Sweden